CLINICAL TRIAL: NCT04586244
Title: An Open-Label, Randomized, Phase 2, Umbrella Study to Investigate the Biological Rational of Various Neoadjuvant Therapies for Participants With Muscle-Invasive Urothelial Carcinoma of the Bladder Who Are Cisplatin-Ineligible or Refuse Cisplatin Therapy and Undergoing Radical Cystectomy
Brief Title: An Umbrella Study to Determine the Safety and Efficacy of Various Monotherapy or Combination Therapies in Neoadjuvant Urothelial Carcinoma
Acronym: Optimus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision. No safety concerns contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-901; 2020-002244-23 (EudraCT Number)
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Urothelial Carcinoma
Keywords: Muscle-invasive cisplatin-ineligible; urothelial carcinoma of the bladder; radical cystectomy.; epacadostat; retifanlimab; TIM-3; LAG-3
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — epacadostat

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment Group A (Experimental): epacadostat will be administered in combination with retifanlimab.
  Interventions: Drug: retifanlimab; Drug: epacadostat
- Treatment Group B (Experimental): retifanlimab will be administered as monotherapy.
  Interventions: Drug: retifanlimab
- Treatment Group C (Experimental): epacadostat will be administered as monotherapy.
  Interventions: Drug: epacadostat
- Treatment Group D (Experimental): retifanlimab will be administered in combination with INCAGN02385.
  Interventions: Drug: retifanlimab; Drug: INCAGN02385
- Treatment Group E (Experimental): retifanlimab will be administered in combination with INCAGN02385 and INCAGN02390.
  Interventions: Drug: retifanlimab; Drug: INCAGN02385; Drug: INCAGN02390

INTERVENTIONS:
Drug: retifanlimab — retifanlimab will be administered via IV over 30 minutes (+ 15 min) on Day 1 of each 28-day cycle, up to 3 cycles,
  Arms: Treatment Group A; Treatment Group B; Treatment Group D; Treatment Group E
Drug: epacadostat — epacadostat will be administered daily twice daily orally up to and including day of surgery.
  Arms: Treatment Group A; Treatment Group C
Drug: INCAGN02385 — INCAGN02385 will be administered via IV over 30 minutes (-5/+10 min) every 2 weeks.
  Arms: Treatment Group D; Treatment Group E
Drug: INCAGN02390 — INCAGN02390 will be administered via IV over 30 minutes (-5/+10 min) every 2 weeks.
  Arms: Treatment Group E

SUMMARY:
This is a multicenter, open-label, randomized, Phase 2 umbrella study of various neoadjuvant treatment combinations in participants who have muscle-invasive urothelial carcinoma of the bladder and are cisplatin-ineligible or refusing cisplatin therapy and awaiting radical cystectomy.

DETAILED DESCRIPTION:
Participants will be stratified based on Programmed cell Death-Ligand 1 (PD-L1) Combined Positive Score ( CPS) < 10 and PD-L1 CPS ≥ 10.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed transitional cell urothelial carcinoma. Participants with mixed histologies are required to have a dominant (ie, 50% at least) transitional cell pattern.
* Clinical stage T2-T3b, N0, M0 muscle invasive urothelial carcinoma by CT (or MRI) (Stage II-IIIA per AJCC 2018)
* Refuse cisplatin therapy (does not apply in France) or are ineligible for cisplatin therapy per modified Galsky criteria with exclusion of Eastern Cooperative Oncology Group( ECOG) PS 2 participants
* Eligible for radical cystectomy
* Eastern Cooperative Oncology Group (ECOG) Performance Status( PS) 0 or 1.
* Pretreatment tumor biopsy must be a tumor block or 20 unstained slides from biopsy of primary tumor containing at least 20% tumor.
* Willingness to avoid pregnancy or fathering children from screening through 100 days in the US and 190 days in Europe after the last dose of study drug

Exclusion Criteria:

* Participation in any other study in which receipt of an investigational study drug or device occurred within 28 days or 5 half-lives (whichever is longer) before first dose.
* Previously received systemic therapy for bladder cancer or received prior treatment with checkpoint inhibitor agents (such as anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4).
* Evidence of measurable nodal or metastatic disease.
* Concurrent anticancer therapy.
* Has had major surgery within 4 weeks before enrollment (C1D1).
* Has had known additional malignancy other than muscle-invasive Urothelial Bladder Cancer ( miUBC) that is progressing or requires active treatment, along with some protocol exceptions, or history of other malignancy within 2 years of study entry, with some predefined-protocol exceptions.
* Has active autoimmune disease requiring systemic immunosuppression with corticosteroids (> 10 mg daily doses of prednisone or equivalent) or immunosuppressive drugs within 2 years of Day 1 of study treatment.
* Participants with laboratory values outside of protocol defined ranges.
* Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg/day of prednisone or equivalent).
* Has a known active hepatitis B (defined as HBsAg and total anti-HBc positive results) or hepatitis C (HCV Ab positive result and HCV RNA >LLoD) or HIV,HBV, HCV or hepatitis virus coinfection.
* Participants with HIV+ disease along with protocol defined exceptions that don't have undetectable viral load along with other protocol exceptions.
* Has known carcinomatous meningitis.
* Active infection requiring systemic antibiotics ≤ 14 days from first dose of study drug.
* Participants with known or suspected active COVID-19 infection.
* Use of probiotics within 28 days from first dose of study drug.
* Current use of prohibited medication as per protocol.
* Has not recovered to ≤ Grade 1 from toxic effects of previous therapy and/or complications from previous surgical intervention.
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically meaningful. A screening QTcF interval > 450 milliseconds is excluded.
* History of a gastrointestinal condition (eg, inflammatory bowel disease, Crohn's disease, ulcerative colitis) that may affect oral drug absorption.
* Has received a live vaccine within 30days of planned start of study therapy
* Participants with impaired cardiac function or clinically significant cardiac disease
* Prior allogenic tissue/solid organ transplant
* Evidence of interstitial lung disease or active, noninfectious pneumonitis.
* Has known hypersensitivity to any of the study drugs, excipients, including mannitol or another monoclonal antibody which cannot be controlled with standard measures (eg, antihistamines and corticosteroids).
* Any ≥ Grade 2 immune-related toxicity while receiving prior immunotherapy.
* History of serotonin syndrome after receiving 1 or more serotonergic drugs.
* Concomitant use of medications that are known to be substrates of CYP1A2, CYP2C8, or CYP2C19 with narrow therapeutic window are prohibited (see Section 6.6.3).
* Patients who are receiving or required to receive medications that are known to be UGT1A9 inhibitors (see Section 6.6.3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Hershock, MD, Study Director — Incyte Corporation
Locations (12):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Medical Center Division of H, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
- France (3):
  - Hopital Europeen Georges Pompidou (Hegp), Paris
  - Hospital Saint Louis, Paris
  - Institut Gustave Roussy, Villejuif
- Italy (5):
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - L Azienda Ospedaliero-Universitaria Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) Ospedale San Raffaele, Milan
  - Universita Campus Bio Medico Di Roma, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma), Verona

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at 2 study centers in the United States, 2 study centers in Italy, and 1 study center in France.
Groups:
- Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W: Participants received oral epacadostat 600 milligrams (mg) twice daily (BID) + intravenous retifanlimab 500 mg every 4 weeks (Q4W; on Day 1 of each 28-day cycle). Treatment continued for 4 to 10 weeks, as long as participants did not meet any criteria for study withdrawal.
- Retifanlimab 500 mg Q4W: Participants received intravenous retifanlimab 500 mg Q4W (on Day 1 of each 28-day cycle). Treatment continued for 4 to 10 weeks, as long as participants did not meet any criteria for study withdrawal.
- Epacadostat 600 mg BID: Participants received oral epacadostat 600 mg BID. Treatment continued for 4 to 10 weeks, as long as participants did not meet any criteria for study withdrawal.
- Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W: Participants received intravenous retifanlimab 500 mg Q4W (on Day 1 of each 28-day cycle) + intravenous INCAGN02385 350 mg every 2 weeks (Q2W). Treatment continued for 4 to 10 weeks, as long as participants did not meet any criteria for study withdrawal.
- Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W: Participants received intravenous retifanlimab 500 mg Q4W (on Day 1 of each 28-day cycle) + intravenous INCAGN02385 350 mg Q2W + intravenous INCAGN02390 400 mg Q2W. Treatment continued for 4 to 10 weeks, as long as participants did not meet any criteria for study withdrawal.
Period: Overall Study
Arm/Group | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W | Retifanlimab 500 mg Q4W | Epacadostat 600 mg BID | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W
Started | 3 | 20 | 2 | 4 | 1
Completed | 2 | 19 | 2 | 3 | 1
Not Completed | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0
Not completed — Surgery Delayed 140 Days Post-Last Dose Due to AE; Follow-up Data Not Collected | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W | Retifanlimab 500 mg Q4W | Epacadostat 600 mg BID | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W | Total
Number analyzed (Participants) | 3 | 20 | 2 | 4 | 1 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (6.66) | 71.1 (6.08) | 65.0 (1.41) | 69.3 (3.86) | NA (NA) — Mean (SD) age cannot be reported for a single participant due to privacy concerns. | NA (NA) — Mean (SD) cannot be reported because doing so would allow for the calculation of the age of the single participant in the retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W arm.
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 1 | 0 | 4
  Male | 3 | 18 | 1 | 3 | 0 | 25
  Cannot Be Reported Due to Participant Privacy | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 2 | 16 | 2 | 4 | 0 | 24
  Not Reported | 1 | 4 | 0 | 0 | 0 | 5
  Cannot Be Reported Due to Participant Privacy | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 15 | 1 | 4 | 0 | 22
  Not Reported | 1 | 5 | 1 | 0 | 0 | 7
  Cannot Be Reported Due to Participant Privacy | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in CD8+ Lymphocytes Within the Resected Tumor
Description: Fold Change from Baseline in CD8+ lymphocytes = CD8+ Lymphocytes at cystectomy divided by CD8+ lymphocytes at Screening. Translational data in all but the retifanlimab 500 mg Q4W treatment group were limited and insufficient to assess this outcome measure.
Time Frame: up to 69 days
Population: Translation Evaluable Population: all participants who enrolled in the study who received at least 4 weeks of neoadjuvant study treatment (needed to receive the last dose of epacadostat within 2 days prior to the day of surgery or needed to receive the last dose of retifanlimab and/or INCAGN02385 and/or INCAGN02390 within the 7 weeks prior to day of surgery) and provided evaluable paired biopsies (pretreatment core biopsy and surgical resection biopsy)
Measure: Mean (Standard Deviation); unit: log 2 of fold change
Arm/Group | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W | Retifanlimab 500 mg Q4W | Epacadostat 600 mg BID | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W
Number analyzed (Participants) | 0 | 6 | 0 | 0 | 0
log 2 of fold change |  | 0.791 (0.9332) |  |  |
Statistical Analysis 1: Comparison: Retifanlimab 500 mg Q4W; Test type: Superiority; p = 0.0925, paired t-test; The paired t-test used n-1 degrees of freedom, where n is the number of evaluable paired samples

2. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as an AE that was reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to 159 days
Population: Safety Population: all participants who received at least 1 dose of study treatment. Treatment groups were determined according to the actual treatment the participant received regardless of the assigned study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W | Retifanlimab 500 mg Q4W | Epacadostat 600 mg BID | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W
Number analyzed (Participants) | 3 | 20 | 2 | 4 | 1
Participants | 3 | 18 | 2 | 4 | 1

3. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. A TEAE was defined as an AE that was reported for the first time or the worsening of a pre-existing event after the first dose of study drug. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5 Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 159 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W | Retifanlimab 500 mg Q4W | Epacadostat 600 mg BID | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W
Number analyzed (Participants) | 3 | 20 | 2 | 4 | 1
Participants | 2 | 9 | 0 | 2 | 1

4. Secondary Outcome: Pathological Complete Response Rate
Description: Pathological complete response rate was defined as the percentage of participants with ypT0N0.
Time Frame: up to 69 days
Population: Efficacy Population: all participants with secondary efficacy endpoint data available for both Baseline and post-Baseline measurements. The 80% confidence interval was estimated using the Clopper-Pearson method.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W | Retifanlimab 500 mg Q4W | Epacadostat 600 mg BID | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W
Number analyzed (Participants) | 2 | 20 | 2 | 4 | 1
percentage of participants | 100 [31.62 to 100] | 40 [24.91 to 56.73] | 0 [0 to 68.38] | 0 [0 to 43.77] | 100 [10 to 100]

5. Secondary Outcome: Major Pathological Response
Description: Major pathological response was defined as the percentage of participants with residual ypT0/1/a/isN0M0.
Time Frame: up to 69 days
Population: Efficacy Population. The 80% confidence interval was estimated using the Clopper-Pearson method.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W | Retifanlimab 500 mg Q4W | Epacadostat 600 mg BID | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W
Number analyzed (Participants) | 2 | 20 | 2 | 4 | 1
percentage of participants | 100 [31.62 to 100] | 50 [33.82 to 66.18] | 50 [5.13 to 94.87] | 50 [14.26 to 85.74] | 100 [10 to 100]

ADVERSE EVENTS:
Time Frame: up to 159 days
Description: Adverse events have been reported for members of the Safety Population, comprised of all participants who received at least 1 dose of study treatment.
Arm/Group | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W | Retifanlimab 500 mg Q4W | Epacadostat 600 mg BID | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/20 | 0/2 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/20 | 0/2 | 1/4 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 18/20 | 2/2 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W (N=3) | Retifanlimab 500 mg Q4W (N=20) | Epacadostat 600 mg BID (N=2) | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W (N=4) | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W (N=1)
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Purulent discharge (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epacadostat 600 mg BID + Retifanlimab 500 mg Q4W (N=3) | Retifanlimab 500 mg Q4W (N=20) | Epacadostat 600 mg BID (N=2) | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W (N=4) | Retifanlimab 500 mg Q4W + INCAGN02385 350 mg Q2W + INCAGN02390 400 mg Q2W (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 3 | 0 | 3 | 0
Hyperpyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 5 | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 1 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0
Carbon dioxide increased (Investigations) | 0 | 0 | 0 | 1 | 0
Inflammatory marker increased (Investigations) | 0 | 2 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Epididymal tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 4 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The sponsor made a strategic decision to stop further enrollment of participants in cohorts encompassing epacadostat in clinical studies. The sponsor later made a strategic decision (not based on safety concerns) to stop enrollment in all treatment groups, and the study was subsequently terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT04586244/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT04586244/SAP_001.pdf